CLINICAL TRIAL: NCT05384067
Title: Defining Stress and Sleep as Modifiable Intervention Targets in Correctional Officers to Reduce Mental and Physical Health Risk
Brief Title: Project MiCRIM- Sleep and Stress Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Scott Pickett, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002715
Record Dates: First submitted 2022-05-12; First posted 2022-05-20 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Sleep; Stress
Keywords: mindfulness; sleep; stress

STUDY DESIGN:
Intervention Model Description: Intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based intervention (Experimental): Participants in this arm will wear a sleep-monitoring device, complete questionnaires and participate in an online mindfulness component each week for the duration of this study.
  Interventions: Behavioral: Mindfulness-based intervention
- Control (No Intervention): Participants in this arm will only wear a sleep-monitoring device and complete questionnaires.

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — Participants will complete one mindfulness education module every week for 4 weeks, and to practice a 15-minute formal guided mindfulness meditation at least five times per week across the 4 weeks. Participants will also be taught evidence-based sleep improvement techniques, will be provided education for when to use the techniques, and will be encouraged to implement the techniques to improve sleep.
  Arms: Mindfulness-based intervention

SUMMARY:
The purpose of Project MiCRIM is to test the feasibility and effectiveness of an online 4-week mindfulness-based intervention that incorporates informational elements about sleep, mindfulness, thoughts, emotions, and acceptance using a control sample of Criminology and Criminal Justice majors as a proxy for Corrections officers.

DETAILED DESCRIPTION:
The study will use a waitlist-control design to examine the effectiveness of a brief (4-week) online mindfulness-based intervention aimed at reducing stress and improving sleep quality. A proxy, convenience sample of 50 criminology majors will be recruited and randomized into the active intervention or waitlist condition. The intervention requires participants to complete one mindfulness education module every week for 4 weeks, and to practice a 15-minute formal guided mindfulness meditation at least five times per week across the 4 weeks. Participants will also be taught evidence-based sleep improvement techniques, will be provided education for when to use the techniques, and will be encouraged to implement the techniques to improve sleep. Validated self-report measures of stress, anxiety, mood, and sleep quality will be assessed pre- and post-intervention. Adherence to the mindfulness practice will be monitored online and self-report assessments of sleep technique implementation will be collected. Sleep patterns will be assessed using a Philips Respironics Spectrum 2 Actiwatch, which is a wrist-worn device that measures movement and light exposure and estimates sleep-wake patterns. Lastly, multiple saliva samples pre- and post-intervention will be collected and analyzed by ELISA with a multiplex cytokine assay. Cortisol, α-amylase, and the four analytes with known deleterious roles in cellular and behavioral stress responsiveness will be measured simultaneously: interleukin-1beta, interleukin-6, interleukin-8, and Tumour Necrosis Factor-alpha will be examined pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

-Criminal Justice or Criminology major

Exclusion Criteria:

* Abnormal BMI (below 18.5 or above 30)
* self-reported sleep apnea, head injury, neurological problem, unstable mental health disorder, substance use disorder, psychosis, or current suicidal ideation or plan

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Saliva Samples via ELISA Assay- Cortisol | Change from baseline to 5 weeks
  Tests for level changes in cortisol.
Saliva Samples via ELISA Assay- α-amylase | Change from baseline to 5 weeks
  Test for level changes in α-amylase.
Saliva Samples via ELISA Assay- interleukin-1beta | Change from baseline to 5 weeks
  Test for level changes in interleukin-1beta.
Saliva Samples via ELISA Assay- interleukin-6 | Change from baseline to 5 weeks
  Test for level changes in interleukin-6.
Saliva Samples via ELISA Assay- interleukin-8 | Change from baseline to 5 weeks
  Test for level changes in interleukin-8.
Saliva Samples via ELISA Assay- TNF-α | Change from baseline to 5 weeks
  Test for level changes in TNF-α.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline to 5 weeks
  Assesses sleep quality. The PSQI includes a scoring key for calculating a patient's seven sub scores, each of which can range from 0 to 3. The sub scores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Pittsburgh Sleep Quality Index, Addendum for PTSD (PSQI-A) | Change from baseline to 5 weeks
  Assesses sleep quality related to PTSD. The PSQI-A includes a scoring key for calculating a patient's scores, each of which can range from 0 to 3 with higher scores indicating worse outcomes.
The Smith Relaxation Dispositions Inventory | Change from baseline to 5 weeks
  Assesses momentary states of relaxation during the past two weeks. Items scored on a 4-point Likert Type scale ranging from 1 (not at all) to 4 (very much).
Five Facet Mindfulness Questionnaire - Short Form | Change from baseline to 5 weeks
  Assesses 5 facets of mindfulness- observation, description, awareness of actions, non-judgement and non-reaction. Items scored on a 5-point Likert-type scale ranging from 1 (never or very rarely true) to 5 (very often or always true). Facet scores were computed by summing the scores on the individual items. Facet scores range from 8 to 40 (except for the nonreactivity facet, which ranges from 7 to 35), with higher scores indicating more mindfulness.
Patient Health Questionnaire 9 | Change from baseline to 5 weeks
  Measures depression severity. This is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 0- not at all, 1- several days, 2- more than half the days, 3- nearly every day, respectively. The total score for the nine items ranges from 0 to 27. 1-4 minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-27 severe depression.
Generalized Anxiety Disorder 7 | Change from baseline to 5 weeks
  Assesses anxiety symptoms. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity. Scores above 10 are considered to be in the clinical range.
Perceived Stress Scale | Change from baseline to 5 weeks
  Assesses perceptions of stress. Scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items.
Sleep Condition Indicator | Change from baseline to 5 weeks
  Eight-item rating scale that was developed to screen for insomnia disorder based on DSM-5 criteria.
The PTSD Checklist for DSM-5 (PCL-5) | Change from baseline to 5 weeks
  Assesses the 20 Diagnostic Statistical Manual-5 symptoms of PTSD using a 5-point Likert-type scale ranging from 0 (not at all) to 4 (extremely).

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University Center for Translational Behavioral Medicine, Tallahassee, Florida, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT05384067/ICF_000.pdf